CLINICAL TRIAL: NCT00284856
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group 6-Month Study to Evaluate the Efficacy and Safety of Oral Montelukast Sodium, Fluticasone Propionate and Placebo in Patients With Chronic Asthma Who Smoke Cigarettes
Brief Title: Montelukast Asthmatic Smoker Study (0476-332)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-332; 2005_108
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Arm 1: Montelukast
  Interventions: Drug: montelukast sodium; Drug: Comparator: Placebo
- 2 (Active Comparator): Arm 2: Fluticasone
  Interventions: Drug: Comparator: fluticasone; Drug: Comparator: Placebo
- 3 (Placebo Comparator): Arm 3: Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: montelukast sodium — montelukast 10 mg tablet once daily, 6 month treatment period
  Arms: 1
Drug: Comparator: Placebo — fluticasone propionate 250 mcg Placebo (Pbo) twice daily, 6 month treatment period
  Arms: 1; 3
Drug: Comparator: fluticasone — fluticasone propionate 250 mcg twice daily, 6 month treatment period
  Arms: 2
Drug: Comparator: Placebo — montelukast 10 mg Pbo tablet once daily, 6 month treatment period
  Arms: 2; 3

SUMMARY:
This is a multicenter study to evaluate the efficacy and safety of MK0476 versus placebo in participants with chronic asthma who actively smoke cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic asthma who actively smoke at least 0.5 to no more than 2 packs of cigarettes a day

Exclusion Criteria:

* Participant cannot have a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) or emphysema.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1640 (Actual)
Dates: Start 2006-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Price D, Popov TA, Bjermer L, Lu S, Petrovic R, Vandormael K, Mehta A, Strus JD, Polos PG, Philip G. Effect of montelukast for treatment of asthma in cigarette smokers. J Allergy Clin Immunol. 2013 Mar;131(3):763-71. doi: 10.1016/j.jaci.2012.12.673. Epub 2013 Feb 4. PMID 23380218

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1640 participants enrolled in the study, 621 participants were excluded during screening and not randomized. The remaining 1019 participants were randomized.
Groups:
- Montelukast: Montelukast 10 mg tablet once daily at bedtime and Fluticasone propionate matching placebo 250 mcg twice daily for 6 months
- Fluticasone: Fluticasone propionate 250 mcg twice daily and Montelukast matching placebo 10 mg tablet once daily at bedtime for 6 months
- Placebo: Montelukast matching placebo 10 mg tablet once daily at bedtime and Fluticasone propionate matching placebo 250 mcg twice daily for 6 months
Period: Overall Study
Arm/Group | Montelukast | Fluticasone | Placebo
Started | 347 | 336 | 336
Completed | 296 | 286 | 276
Not Completed | 51 | 50 | 60
Not completed — Adverse Event | 3 | 3 | 3
Not completed — Lack of Efficacy | 2 | 1 | 8
Not completed — Lost to Follow-up | 25 | 21 | 22
Not completed — Protocol Violation | 5 | 4 | 5
Not completed — Withdrawal by Subject | 12 | 16 | 18
Not completed — Other | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast | Fluticasone | Placebo | Total
Number analyzed (Participants) | 347 | 336 | 336 | 1019
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.4) | 38.4 (10.7) | 37.9 (9.9) | 38.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 147 | 166 | 476
  Male | 184 | 189 | 170 | 543

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Asthma-control Days Over the 6-month Treatment Period
Description: An asthma-control day, computed from daily diaries, was any day with no unscheduled visit for asthma care, no use of > than 2 puffs of β-agonist, no use of other asthma rescue medication, and no nocturnal awakening. The percentage of asthma-control days was the number of days with asthma-control divided by the total number of days with non-missing values for this endpoint. The patient diary had questions concerning daytime and nighttime symptoms, morning (AM) and evening (PM) peak expiratory flow rate (PEFR), β-agonist use, asthma attacks and smoking activity.
Time Frame: 6 months
Population: Efficacy analysis was based on the full analysis set (FAS) population which included all participants who had at least 7 days of on-treatment data for the specific endpoint. Thirty three patients were excluded from the FAS (13 on montelukast, 7 on fluticasone and 13 on placebo). One participant in the placebo group did not take study medication.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Montelukast | Fluticasone | Placebo
Number analyzed (Participants) | 334 | 329 | 323
Percentage of days | 50.70 (38.19) [40.62 to 49.33] | 53.30 (39.06) [44.86 to 53.53] | 43.84 (38.08) [34.65 to 43.45]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; Least Squares Mean Difference = 5.92, 95% CI [0.28 to 11.56] — Estimated Value is difference in least squares mean (montelukast - placebo)
Statistical Analysis 2: Comparison: Fluticasone vs Placebo; Test type: Superiority or Other; Least Squares Mean Difference = 10.14, 95% CI [4.50 to 15.78] — Estimated value is difference in least squares mean (fluticasone - placebo)
Statistical Analysis 3: Comparison: Montelukast vs Fluticasone; Test type: Superiority or Other; Least Squares Mean Difference = -4.22, 95% CI [-9.83 to 1.38] — Estimated value is difference in least squares mean (montelukast - fluticasone)

2. Secondary Outcome: Change From Baseline in Mean Daytime Symptom Score Over a 6-month Treatment Period
Description: 4 daytime symptoms were evaluated daily on a 7-point scale from 0 (best)- 6 (worst). The on-treatment daytime symptom score was computed by averaging over Period II the mean of the 4 daily symptom scores recorded daily in the diary while the baseline daytime symptom score was obtained by averaging the mean of the 4 daily symptom scores across the daily diary entries of the Baseline period (Period I). The change from baseline in mean daytime symptom score is computed as the difference between the mean on-treatment daytime symptom score & the mean baseline daytime symptom score.
Time Frame: Baseline and 6 months
Population: Efficacy analysis was based on the full analysis set (FAS) population which included all participants who received at least one dose of the randomized double-blind study medication and who had at least 7 days of on-treatment data for the specific endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Montelukast | Fluticasone | Placebo
Number analyzed (Participants) | 335 | 329 | 322
Score on a scale
  Baseline | 1.82 (1.03) [-0.53 to -0.37] | 1.78 (0.97) [-0.58 to -0.42] | 1.90 (0.94) [-0.38 to -0.23]
  Average Change from Baseline During Period II | -0.41 (0.70) | -0.44 (0.68) | -0.27 (0.72)
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; Least Squares Mean Difference = -0.15, 95% CI [-0.25 to -0.05] — Estimated value is difference in least squares mean (montelukast - placebo)
Statistical Analysis 2: Comparison: Fluticasone vs Placebo; Test type: Superiority or Other; Least Squares Mean Difference = -0.20, 95% CI [-0.30 to -0.10] — Estimated value is difference in least squares mean (fluticasone - placebo)
Statistical Analysis 3: Comparison: Montelukast vs Fluticasone; Test type: Superiority or Other; Least Squares Mean Difference = 0.05, 95% CI [-0.05 to 0.15] — Estimated value is difference in least squares mean (montelukast - fluticasone)

3. Secondary Outcome: Change From Baseline in Average Morning (AM) PEFR (Peak Expiratory Flow Rate) Over a 6-month Treatment Period
Description: PEFR measurements were performed daily, in the morning before using any medication. The on-treatment AM PEFR was computed by averaging over Period II (treatment period) the AM PEFR recorded daily in the diary, while the baseline AM PEFR was obtained by averaging the AM PEFR across the daily diary entries of the Baseline Period or Period I (placebo run-in period). The change from baseline in average AM PEFR is computed as the difference between mean on-treatment AM PEFR and mean baseline AM PEFR.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Montelukast | Fluticasone | Placebo
Number analyzed (Participants) | 334 | 329 | 324
Liters/minute
  Baseline | 363.75 (112.40) | 354.28 (101.64) | 347.98 (99.21)
  Average Change from Baseline During Period II | 12.84 (40.22) | 19.31 (44.85) | 8.27 (40.70)
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; Least Squares Mean Difference = 5.09, 95% CI [-1.27 to 11.45] — Estimated value is difference in least squares mean (montelukast - placebo)
Statistical Analysis 2: Comparison: Fluticasone vs Placebo; Test type: Superiority or Other; Least Squares Mean Difference = 11.21, 95% CI [4.85 to 17.58] — Estimated value is difference in least squares mean (fluticasone - placebo)
Statistical Analysis 3: Comparison: Montelukast vs Fluticasone; Test type: Superiority or Other; Least Squares Mean Difference = -6.13, 95% CI [-12.46 to 0.20] — Estimated value is difference in least squares mean (montelukast - fluticasone)

ADVERSE EVENTS:
Description: The population for safety analyses was the All Patients as Treated (APaT) set.
  The set included all randomized participants who took at least one dose of the
  double-blind study medication. One participant in the placebo group was randomized but did not take treatment. Therefore, participant was not included in the safety analyses.
Arm/Group | Montelukast | Fluticasone | Placebo
Serious Adverse Events (participants affected / at risk) | 9/347 | 10/336 | 11/335
Other Adverse Events (participants affected / at risk) | 65/347 | 57/336 | 72/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=347) | Fluticasone (N=336) | Placebo (N=335)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Salpingo-oophoritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 6 (7)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5) | 2 (3)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=347) | Fluticasone (N=336) | Placebo (N=335)
Nasopharyngitis (Infections and infestations) | 23 (30) | 27 (34) | 22 (26)
Asthma (Respiratory, thoracic and mediastinal disorders) | 45 (71) | 34 (50) | 57 (95)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts,

manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as

confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.